CLINICAL TRIAL: NCT05573256
Title: Effects of Sleep Hygiene Education and Lavender Oil Inhalation on Sleep Quality, Fatigue, and Health-related Quality of Life in Adults With a Stoma: A Randomized Controlled Trial Protocol
Brief Title: Effects of Sleep Hygiene Education and Lavender Oil Inhalation on Sleep Quality, Fatigue, Quality of Life
Acronym: MU-RKOCA-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: MU-RKOCA-01
Record Dates: First submitted 2022-10-07; First posted 2022-10-10 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Ostomy
Keywords: Ostomy; Sleep Hygiene; Lavander oil; Sleep; Fatigue; Quality of Life
MeSH Terms: conditions — Sleep Hygiene; Fatigue

STUDY DESIGN:
Intervention Model Description: Every night before going to bed (21:00-24:00), the participants will drop two drops of 2% lavender essential oil on a 2x2 cm cotton gauze pad in a bowl, place it at a distance of 15-20 cm from their pillows, and breath normally for 20 minutes. The participants will be instructed to repeat this process by dripping lavender oil onto a new gauze pad every night for four weeks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Sleep hygiene education together with lavender oil inhalation) (Experimental): the participants assigned to Group 1 will be given sleep hygiene education and instructed how to apply lavender oil inhalation. The participants will be provided with charts on sleep hygiene education and lavender oil inhalation and shown how to regularly keep daily records using their charts. The participants in this group will be given a copy of the sleep hygiene education brochure and lavender oil in a 10 ml bottle.
  Interventions: Behavioral: Lavender oil inhalation; Behavioral: Sleep hygiene education
- Group 2 (Sleep hygiene education) (Experimental): The participants assigned to Group 2 will only be given sleep hygiene education. They will be provided with a copy of the sleep hygiene education brochure and a chart on which to record their sleep hygiene practices.
  Interventions: Behavioral: Sleep hygiene education
- Group 3 (Lavender oil inhalation) (Experimental): The participants assigned to Group 3 will only be instructed on how to apply lavender oil inhalation and keep regular daily records on the chart given. The participants in this group will be given lavender oil in a 10 ml bottle.
  Interventions: Behavioral: Lavender oil inhalation
- Group 4 (Routine care) (No Intervention): Participants assigned to Group 4 will be given routine care and no application will be made.
  Patient care and follow-up are routinely performed as follows: Following the patient's admission to the clinic, the first evaluation of the patient is made by the ostomy and wound care nurses within 24 hours, and patient education is initiated accompanied by the primary caregiver from the family. Throughout the period from admission to clinic to discharge, the ostomy care and education of the patient is repeated by the ostomy and wound care nurses every 72 hours. In addition, the patient and caregiver are given the contact information of the ostomy and wound care nurses and informed that they can call them at any time when they need it after discharge from the hospital.

INTERVENTIONS:
Behavioral: Lavender oil inhalation — Lavender oil inhalation;During the trial, the participants will be asked to practice lavender oil inhalation as follows: Every night before going to bed (21:00-24:00), the participants will drop two drops of 2% lavender essential oil on a 2x2 cm cotton gauze pad in a bowl, place it at a distance of 15-20 cm from their pillows, and breath normally for 20 minutes. The participants will be instructed to repeat this process by dripping lavender oil onto a new gauze pad every night for four weeks.
  Arms: Group 1 (Sleep hygiene education together with lavender oil inhalation); Group 3 (Lavender oil inhalation)
Behavioral: Sleep hygiene education — Sleep hygiene education;The participants assigned to Groups 1 and 2 will receive sleep hygiene education using the sleep hygiene education brochure, which has been prepared by the researchers based on the literature concerning the improvement of general sleep quality in individuals with a stoma.
  Arms: Group 1 (Sleep hygiene education together with lavender oil inhalation); Group 2 (Sleep hygiene education)

SUMMARY:
Self-care non-pharmacological methods can help reduce the negative health effects of sleep problems or insomnia. This trial aims to investigate the effects of sleep hygiene education and lavender oil inhalation alone and in combination on sleep quality, fatigue, and health-related quality of life in adults with a stoma.

DETAILED DESCRIPTION:
This study has been planned as a randomized controlled clinical trial and will use a 2x2 factor design in which an equal number of participants meeting the inclusion criteria will be randomly allocated to one of four groups. The study population will comprise 120 adult patients who have undergone ostomy surgery in a city hospital in Turkey. Lavender oil inhalation together with sleep hygiene education will be applied in the first group (n=30), only sleep hygiene education in the second group (n=30), only lavender oil inhalation in the third group (n=30), and no intervention in the fourth group (n=30). The sleep quality of the groups will be evaluated using the Pittsburgh Sleep Quality Index, their fatigue levels with the Chalder Fatigue Scale, and their quality of life with the Stoma Quality of Life Scale.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* At least three months having passed after ostomy,
* Having a clear level of consciousness and no disease or medication use that can negatively affect the level of consciousness,
* Being able to communicate in Turkish,
* Providing informed written consent to participate in the study.

Exclusion Criteria:

* Lavender allergy,
* Respiratory tract infections such as sinusitis and pneumonia,
* Body mass index (BMI) of >40,
* A diagnosis of sleep disorder and/or medication use for sleep problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | a month
  . It consists of seven subscales with a total of 19 items, of which 18 are included in scoring. Each item is evaluated over 0-3 points, and the sum of the seven subscale scores constitutes the total PSQI score. The total score that can be obtained from the scale ranges from 0 to 21, and a high total score indicates poor sleep quality. A total PSQI score of ≤5 indicates 'good sleep', and a score of >5 indicates 'poor sleep'.
Chalder Fatigue Scale (CFS) | a month
  The scale consists of 11 items, seven evaluating physical fatigue and four evaluating mental fatigue. There are four options for response to the items in the scale (less than usual, no more than usual, more than usual, and much more than usual). The overall fatigue score is obtained by summing the scores in the physical and mental fatigue subscales. The physical fatigue subscale score ranges from 0 to 21, the mental fatigue subscale score ranges from 0 to 12, and the total fatigue score ranges from 0 to 33. An increase in the scale score indicates an increase in the severity of fatigue.
Stoma Quality of Life Scale (SQLS) | a month
  The remaining items are grouped into three subscales: work/social life (six items), sexuality/body image (five items), and stoma function (six items). In addition, there is one item related to the economic situation and one item related to skin irritation, which do not fall into any of the previously mentioned subscales. Minimum and maximum scores for each subscale are 0 and 100, respectively, with high scores indicating an increase in quality of life. If two items in any subscale are left unanswered in the scale, the relevant subscale is not taken into consideration during scoring, but if one item is left unanswered, it can be included in evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Koca, Principal Investigator — Marmara University, Institute of Health Sciences
Locations (1):
- Rabia Koca, Istanbul, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambe PC, Kurz NR, Nitschke C, Odeh SF, Moslein G, Zirngibl H. Intestinal Ostomy. Dtsch Arztebl Int. 2018 Mar 16;115(11):182-187. doi: 10.3238/arztebl.2018.0182. PMID 29607805
- [Background] Fingren J, Lindholm E, Petersen C, Hallen AM, Carlsson E. A Prospective, Explorative Study to Assess Adjustment 1 Year After Ostomy Surgery Among Swedish Patients. Ostomy Wound Manage. 2018 Jun;64(6):12-22. PMID 30059344
- [Background] Zhang Y, Xian H, Yang Y, Zhang X, Wang X. Relationship between psychosocial adaptation and health-related quality of life of patients with stoma: A descriptive, cross-sectional study. J Clin Nurs. 2019 Aug;28(15-16):2880-2888. doi: 10.1111/jocn.14876. Epub 2019 May 5. PMID 30939212
- [Background] Temiz Z, Cavdar I, Ozbas A, Altunsoy M, Akyuz N, Kutlu FY. Sleep Quality and Factors Affecting Sleep in Individuals With an Intestinal Ostomy: A Descriptive Cross-Sectional Study. Wound Manag Prev. 2022 May;68(5):28-36. doi: 10.25270/wmp.2022.5.2836. PMID 35617011
- [Background] Pachler J, Wille-Jorgensen P. Quality of life after rectal resection for cancer, with or without permanent colostomy. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD004323. doi: 10.1002/14651858.CD004323.pub4. PMID 23235607
- [Background] Krouse R, Grant M, Ferrell B, Dean G, Nelson R, Chu D. Quality of life outcomes in 599 cancer and non-cancer patients with colostomies. J Surg Res. 2007 Mar;138(1):79-87. doi: 10.1016/j.jss.2006.04.033. Epub 2006 Dec 29. PMID 17196990
- [Background] Cavdar I, Temiz Z, Ozbas A, Can G, Tarhan F, Findik UY, Kutlu FY, Akyuz N. Sleep and quality of life in people with ileal conduit. Scand J Urol. 2016 Dec;50(6):472-476. doi: 10.1080/21681805.2016.1236834. Epub 2016 Oct 5. PMID 27701970
- [Background] Carlsson E, Berglund B, Nordgren S. Living with an ostomy and short bowel syndrome: practical aspects and impact on daily life. J Wound Ostomy Continence Nurs. 2001 Mar;28(2):96-105. doi: 10.1067/mjw.2001.113261. PMID 11248730
- [Background] Vorbeck E, Willette-Murphy K, Meiers S, Rudel R, Alakhras M. A descriptive study to assess the impact of surgical stomas on individuals' sleep perceptions & response to sleep hygiene. Ostomy Wound Manage. 2010 Jan 1;56(1):36-44. PMID 20093716
- [Background] Baldwin CM, Grant M, Wendel C, Hornbrook MC, Herrinton LJ, McMullen C, Krouse RS. Gender differences in sleep disruption and fatigue on quality of life among persons with ostomies. J Clin Sleep Med. 2009 Aug 15;5(4):335-43. PMID 19968011
- [Background] Furukawa C, Morioka I. Health-Related Quality of Life and Sleep Disorders in Patients With a Urostomy: Is There a Relationship? J Wound Ostomy Continence Nurs. 2017 Jul/Aug;44(4):358-362. doi: 10.1097/WON.0000000000000334. PMID 28549047
- [Background] Lillehei AS, Halcon LL, Savik K, Reis R. Effect of Inhaled Lavender and Sleep Hygiene on Self-Reported Sleep Issues: A Randomized Controlled Trial. J Altern Complement Med. 2015 Jul;21(7):430-8. doi: 10.1089/acm.2014.0327. Epub 2015 Jun 2. PMID 26133206
- [Background] Stepanski EJ, Wyatt JK. Use of sleep hygiene in the treatment of insomnia. Sleep Med Rev. 2003 Jun;7(3):215-25. doi: 10.1053/smrv.2001.0246. PMID 12927121
- [Background] Lytle J, Mwatha C, Davis KK. Effect of lavender aromatherapy on vital signs and perceived quality of sleep in the intermediate care unit: a pilot study. Am J Crit Care. 2014 Jan;23(1):24-9. doi: 10.4037/ajcc2014958. PMID 24382614
- [Background] van der Ploeg ES, Eppingstall B, O'Connor DW. The study protocol of a blinded randomised-controlled cross-over trial of lavender oil as a treatment of behavioural symptoms in dementia. BMC Geriatr. 2010 Jul 22;10:49. doi: 10.1186/1471-2318-10-49. PMID 20649945
- [Background] Cho MY, Min ES, Hur MH, Lee MS. Effects of aromatherapy on the anxiety, vital signs, and sleep quality of percutaneous coronary intervention patients in intensive care units. Evid Based Complement Alternat Med. 2013;2013:381381. doi: 10.1155/2013/381381. Epub 2013 Feb 17. PMID 23476690
- [Background] van der Watt G, Janca A. Aromatherapy in nursing and mental health care. Contemp Nurse. 2008 Aug;30(1):69-75. doi: 10.5172/conu.673.30.1.69. PMID 19072192
- [Background] Karadag E, Samancioglu S, Ozden D, Bakir E. Effects of aromatherapy on sleep quality and anxiety of patients. Nurs Crit Care. 2017 Mar;22(2):105-112. doi: 10.1111/nicc.12198. Epub 2015 Jul 27. PMID 26211735
- [Background] Ayik C, Ozden D. The effects of preoperative aromatherapy massage on anxiety and sleep quality of colorectal surgery patients: A randomized controlled study. Complement Ther Med. 2018 Feb;36:93-99. doi: 10.1016/j.ctim.2017.12.002. Epub 2017 Dec 6. PMID 29458940
- [Background] Muz G, Tasci S. Effect of aromatherapy via inhalation on the sleep quality and fatigue level in people undergoing hemodialysis. Appl Nurs Res. 2017 Oct;37:28-35. doi: 10.1016/j.apnr.2017.07.004. Epub 2017 Aug 1. PMID 28985917
- [Background] Genc F, Karadag S, Kilic Akca N, Tan M, Cerit D. The Effect of Aromatherapy on Sleep Quality and Fatigue Level of the Elderly: A Randomized Controlled Study. Holist Nurs Pract. 2020 May/Jun;34(3):155-162. doi: 10.1097/HNP.0000000000000385. PMID 32282491
- [Background] Hamzeh S, Safari-Faramani R, Khatony A. Effects of Aromatherapy with Lavender and Peppermint Essential Oils on the Sleep Quality of Cancer Patients: A Randomized Controlled Trial. Evid Based Complement Alternat Med. 2020 Mar 25;2020:7480204. doi: 10.1155/2020/7480204. eCollection 2020. PMID 32308715
- [Background] Bakhtiari S, Paki S, Khalili A, Baradaranfard F, Mosleh S, Jokar M. Effect of lavender aromatherapy through inhalation on quality of life among postmenopausal women covered by a governmental health center in Isfahan, Iran: A single-blind clinical trial. Complement Ther Clin Pract. 2019 Feb;34:46-50. doi: 10.1016/j.ctcp.2018.11.001. Epub 2018 Nov 7. PMID 30712745
- [Background] Berti-Hearn L, Elliott B. Colostomy Care: A Guide for Home Care Clinicians. Home Healthc Now. 2019 Mar/Apr;37(2):68-78. doi: 10.1097/NHH.0000000000000735. PMID 30829784
- [Background] Cengiz B, Bahar Z. Perceived Barriers and Home Care Needs When Adapting to a Fecal Ostomy: A Phenomenological Study. J Wound Ostomy Continence Nurs. 2017 Jan/Feb;44(1):63-68. doi: 10.1097/WON.0000000000000271. PMID 27564927
- [Background] Taylor C, Munro J, Goodman W, Beeken RJ, Dames N, Oliphant R, Watson AJ, Hubbard G. Experiences of wearing support garments by people living with a urostomy. Br J Nurs. 2019 Dec 12;28(22):S26-S33. doi: 10.12968/bjon.2019.28.22.S26. PMID 31835944
- [Background] Lim SH, Chan SW, He HG. Patients' Experiences of Performing Self-care of Stomas in the Initial Postoperative Period. Cancer Nurs. 2015 May-Jun;38(3):185-93. doi: 10.1097/NCC.0000000000000158. PMID 24836957
- [Background] Basch E, Foppa I, Liebowitz R, Nelson J, Smith M, Sollars D, Ulbricht C. Lavender (Lavandula angustifolia Miller). J Herb Pharmacother. 2004;4(2):63-78. PMID 15364646
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Chalder T, Berelowitz G, Pawlikowska T, Watts L, Wessely S, Wright D, Wallace EP. Development of a fatigue scale. J Psychosom Res. 1993;37(2):147-53. doi: 10.1016/0022-3999(93)90081-p. PMID 8463991
- [Background] Baxter NN, Novotny PJ, Jacobson T, Maidl LJ, Sloan J, Young-Fadok TM. A stoma quality of life scale. Dis Colon Rectum. 2006 Feb;49(2):205-12. doi: 10.1007/s10350-005-0275-6. PMID 16392025